CLINICAL TRIAL: NCT05480254
Title: The Effect on Catheter-Related Complıcatıons of Clamping Method the Indwelling Urinary Catheters in ICU Patıents: A Randomızed Controlled Trial
Brief Title: The Effect of Clamping Method the Indwelling Urinary Catheters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hulya Kocyigit (Other)
Collaborators: Cumhuriyet University (Other)
Responsible Party: Sponsor-Investigator, Hulya Kocyigit, Principal Investigator, Cumhuriyet University
Organization: Cumhuriyet University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Cumhuriyet Universty
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Bladder Training by Clamping Before Removal
Keywords: Clamping; Indwelling Urinary Catheters; Nursing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clamped catheter group (Experimental): Q3 clamped catheter protocol is applied before urinary catheter removal
  Interventions: Other: clamped catheter
- free dranaige group (No Intervention): Free dranaige is applied before urinary catheter removal

INTERVENTIONS:
Other: clamped catheter — Q3 clamped catheter protocol is applied before urinary catheter removal
  Arms: clamped catheter group

SUMMARY:
Background: Bladder training through catheter clamping is an important nursing practice. There is no clear information and sufficient evidence for catheter clamping in bladder training before urinary catheter removal in guidelines for clinical practice.

Objective: To evaluate the results of bladder training in ICU patients. Design: Randomized controlled trial. Setting general surgery ıntensıve care. Methods: Patients were randomly assigned either to have their urinary catheter clamped before removal or to have their catheter removed with free drainage.. Patients who will continue to have urinary catheterization for at least 5 days were included in the study.

Results: - Conclusion: -

DETAILED DESCRIPTION:
Nurses are key professionals in the prevention of complications associated with indwelling urinary catheterization in the hospital setting. In this context, bladder training through catheter clamping is an important nursing practice. Indwelling catheter clamping in bladder training was first proposed by Ross in 1936. There is no clear information and sufficient evidence for catheter clamping in bladder training before urinary catheter removal in national and international guidelines for clinical practice.

In a study by Williamson (1982) on this subject, it was reported that intermittent clamping before removal of the indwelling urinary catheter reduces the frequency of urinary retention and shortens the time to return to normal bladder function. However, a systematic review published in Cochrane (2007) on strategies for removal of short-term indwelling urethral catheters in adults found insufficient evidence to suggest that catheter clamping prior to termination of catheterization is effective to induce normal bladder filling. In another systematic review published in Cochrane (2016), there was no significant difference between the patients' subjective perceptions of recatheterization, urinary retention, catheter-related urinary tract infection and urination symptoms in the clamping and free drainage groups.

In the limited number of studies on bladder training performed by clamping the indwelling urinary catheter, no evidence for practice could be obtained, and there is no consensus among clinicians yet. Ultimately, more research, better quality methodology, and more diverse study designs are needed until strong evidence is available to remove this uncertainty.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Scale between 13-15 when clamping will be performed.
* Within the first 12 hours of admission to the intensive care unit,
* Will continue urinary catheterization for at least 5 days,
* No diagnosed or recurrent urinary tract infection,
* Patients who agreed to participate in the study by obtaining their informed consent and who will not leave the study during the study.

Exclusion Criteria:

* Having urinary outflow resistance/difficulty (prostate enlargement, urethral stenosis, etc.),
* Those who have suprapubic catheters or who will undergo intermittent catheterization,
* Patients with impaired nerve conduction,
* Patients taking anticholinergic drug therapy such as tricyclic antidepressants,
* Patients receiving sympathomimetric drug therapy,
* Having a neurogenic bladder,
* Having diabetic cystopathy, Have a previous history of urinary retention or urination dysfunction,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Yes
Enrollment: 110 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Enfectious complications | 1-5 days
  Catheter-Related Infectious Complications Follow-up Form

SECONDARY OUTCOMES:
Other complications | 6. days 1-12 hour between
  Catheter-Related Non-Infectious Complications Follow-up Form

CONTACTS AND LOCATIONS:
Locations (1):
- Cumhuriyet Universty, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will share in 6 months